CLINICAL TRIAL: NCT06652269
Title: The Impact of Equine-Assisted Psychotherapy on Depression, Anxiety, and Stress in Patients with Substance Use Disorder in a Psychiatric Hospital
Status: Completed | Type: Observational
Sponsor: Czech University of Life Sciences Prague (Other)
Responsible Party: Principal Investigator, doc. Ing. Kristýna Machová, Ph.D., Associate professor, Advanced Bionics
Other Study IDs: 8870-VIII/2013
Record Dates: First submitted 2024-10-10; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Substance Abuse Disorder; Anxiety; Depression Secondary to Other Disease
Keywords: Equine asssited psychotherapy; substance use disorder; psychotherapy
MeSH Terms: conditions — Substance-Related Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — Psychometric scales
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental: Group with equine-assisted psychotherapy
  Interventions: Other: Psychopharmacology intervention
- Control: Group with psychotherapy

INTERVENTIONS:
Other: Psychopharmacology intervention — Psychotherapy with horses
  Groups: Experimental

SUMMARY:
This study aims to assess whether an EAP program affects anxiety, depression, and stress, which are often associated with substance use disorder. The management of these conditions has a major impact on the control of the addiction.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of an EAP program on 32 respondents in the experimental group and 36 in the control group. These respondents were patients in a psychiatric hospital who were taking part in an addiction treatment program. The EAP program was conducted weekly over four weeks, with each session lasting three hours. The treatment effects were assessed using the STAI-Y modules 1 and 2, BAI, PSS, and DASS-21 questionnaires. The groups were compared before and after the four-week observation period.

ELIGIBILITY:
Inclusion Criteria:

Patients of psychiatric hospital of Kosmonosy with substance use disorder

Exclusion Criteria:

Exclusion criteria were possible cognitive deficit or reluctance to work with animals. Participants who did not complete all required materials or left the treatment program before completion were excluded from the study (N = 9).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of psychiatric hospital with substance use disorder
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | through study completion, an average of 18 months
  The State-Trait Anxiety Inventory (STAI) is an instrument evaluating the current level of anxiety and personality traits. It was translated into the czech in 2019 by Figalová (2019). Scoring is done using a template, and the range of final scores is 20-80 for each subscale. The higher the score, the higher the level of anxiety or fear. The scores can be divided into three categories-no or low perceived anxiety/anxiousness, moderate anxiety/anxiousness, and high anxiety/anxiousness (Müllner et. al, 1980; Figalová, 2019).
Depression Anxiety and Stress Scale 21 (DASS-21) | through study completion, an average of 18 months
  The DASS-21 scale has 21 items. Respondents rate their experiences in the past week on a four-point Likert scale (0 = not at all; 1 = sometimes; 2 = often; 3 = almost always). The questionnaire has three subscales: depression, anxiety, and stress. The depression subscale focuses on the patient's low mood, anhedonia, hopelessness, self-deprecation, devaluation of life, and decreased motivation. The anxiety subscale focuses on physiological arousal, subjective feelings of tension, situational anxiety, and fear. The stress subscale measures the inability to relax, tension, impatience, and irritability. For all three subscales, scores are categorized as normal, mild, moderate, severe, and extremely severe (Lovibond & Lovibond, 1995).
Perceived Stress Scale (PSS) | through study completion, an average of 18 months
  The Perceived Stress Scale (PSS) is a self-report scale to measure non-specific perceived stress (Cohen et. al, 1983). It is a short scale that is easy to administer, can be administered individually or in groups, is easy to score, and has satisfactory psychometric properties despite its small size. It is the most commonly used psychological instrument to measure perceived stress (Cohen & Janicki-Deverts, 2009). The scale consists of 10 items. Within the PSS, scores can be divided into three categories: low stress, moderate stress, and high perceived stress (Buršíková et al., 2018).
Beck Anxiety Inventory (BAI) | through study completion, an average of 18 months
  The Beck Anxiety Inventory (BAI; [Beck et al., 1988]) is a self-report instrument useful for assessing general anxiety in patients with anxiety disorders or depression. The BAI allows for the assessment of actual levels of anxiety. It assesses the expression of both somatic and psychological symptoms of anxiety. The questionnaire has excellent internal consistency (Cronbach's alpha = 0.92) and satisfactory test-retest performance (r = 0.75) at one week. The categories can be divided into minimal anxiety, mild anxiety, moderate anxiety, and severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Kristýna Machová, associate professor, Principal Investigator — Czech university of life sciences
Locations (1):
- Psychiatrická nemocnice Kosmonosy, Kosmonosy, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All data are available on Mendeley database (10.17632/bng79xc6pc.1).
Supporting Information: Analytic Code
Time Frame: Unending- All data are available on Mendeley database https://data.mendeley.com/datasets/bng79xc6pc/1
Access Criteria: All data are available on Mendeley database https://data.mendeley.com/datasets/bng79xc6pc/1